CLINICAL TRIAL: NCT06314074
Title: Oscillometric Blood Pressure Measurement At 2.5- Vs. 5-minute Intervals and Hypotension in Patients Having Non-cardiac Surgery: a Randomized Trial
Brief Title: 2.5 Versus 5 Minutes Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Karim Kouz, Dr. Karim Kouz, Principal Investigator, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-101143-BO-ff
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-03

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oscillometric blood pressure monitoring at 2.5-minute intervals (Experimental): In patients assigned to oscillometric blood pressure monitoring at 2.5-minute intervals, oscillometric upper-arm cuff blood pressure will be measured and displayed on the patient monitor every 2.5 minutes during surgery.
  Blood pressure will additionally measured with BLINDED continuous non-invasive finger-cuff blood pressure monitoring.
  Interventions: Other: Oscillometric blood pressure monitoring at 2.5-minute intervals
- Oscillometric blood pressure monitoring at 5-minute intervals (Active Comparator): In patients assigned to oscillometric blood pressure monitoring at 5-minute intervals, oscillometric upper-arm cuff blood pressure will be measured and displayed on the patient monitor every 5 minutes during surgery.
  Blood pressure will additionally measured with BLINDED continuous non-invasive finger-cuff blood pressure monitoring.
  Interventions: Other: Oscillometric blood pressure monitoring at 5-minute intervals

INTERVENTIONS:
Other: Oscillometric blood pressure monitoring at 2.5-minute intervals — Oscillometric blood pressure will be measured at 2.5-minute intervals during surgery.
  Arms: Oscillometric blood pressure monitoring at 2.5-minute intervals
Other: Oscillometric blood pressure monitoring at 5-minute intervals — Oscillometric blood pressure will be measured at 5-minute intervals during surgery.
  Arms: Oscillometric blood pressure monitoring at 5-minute intervals

SUMMARY:
This is a randomized trial investigating the effect of oscillometric blood pressure monitoring at 2.5-minute intervals - compared to 5-minute intervals - on intraoperative hypotension. Specifically, the investigators will test the primary hypothesis that oscillometric blood pressure monitoring at 2.5-minute intervals - compared to 5-minute intervals - reduces the time-weighted average mean arterial pressure below 65 mmHg in patients having non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥45 years
* scheduled for elective non-cardiac surgery under general anesthesia
* planned oscillometric blood pressure monitoring with an upper-arm cuff
* American Society of Anesthesiologists physical status class II or higher

Exclusion Criteria:

* emergency surgery
* arm or shoulder surgery
* pregnancy
* preoperative blood pressure differences between the right and left arm of more than 20 mmHg
* intraoperative invasive blood pressure monitoring
* previous preoperative peripheral nerve injury (such as diabetic neuropathy, carpal tunnel syndrome, or cervical radiculopathy)
* contraindication for continuous finger-cuff blood pressure monitoring (e.g., Raynaud's disease, arterial-venous shunts, or cardiac assist devices)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Time-weighted average mean arterial pressure <65 mmHg | Beginning of surgery until the end of surgery
  The primary endpoint will be the time-weighted average mean arterial pressure <65 mmHg (continuous outcome) - defined as the area under a MAP of 65 mmHg divided by the time of continuous finger-cuff blood pressure monitoring [mmHg].

SECONDARY OUTCOMES:
Episodes of a mean arterial pressure <50 mmHg | Beginning of surgery until the end of surgery
  Absolute number of patients with at least one 1-minute episode of a mean arterial pressure <50 mmHg.
Norepinephrine dose | Beginning of surgery until the end of surgery
  Time-weighted cumulative amount of norepinephrine indexed to body weight [µg/kg/min].

CONTACTS AND LOCATIONS:
Overall Officials: Karim Kouz, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany